CLINICAL TRIAL: NCT03008876
Title: The Efficacy of IV Acetaminophen on Patent Ductus Arteriosus Closure in Preterm Infants
Brief Title: IV Acetaminophen and Patent Ductus Arteriosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Kate Tauber, Assistant Professor, Albany Medical College
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4683
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Patent Ductus Arteriosus
Keywords: neonate; acetaminophen
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acetaminophen (Experimental): Group of patients randomized to receive acetaminophen to treat their PDA
  Interventions: Drug: Acetaminophen
- ibuprofen (Active Comparator): Group of patients randomized to receive ibuprofen to treat their PDA
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — infants receive acetaminophen for treatment of their PDA
  Other Names: tylenol
  Arms: acetaminophen
Drug: Ibuprofen — infants receive ibuprofen, standard of care in our unit, for treatment of a PDA
  Arms: ibuprofen

SUMMARY:
This is a randomized controlled trial to evaluate the efficacy of IV acetaminophen versus IV ibuprofen in closing a hemodynamically significant patent ductus arteriosus in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants 23-30 weeks gestation,
* PDA requiring treatment

Exclusion Criteria:

* infection,
* congenital heart disease,
* genetic syndrome,
* NEC,
* pulmonary hypertension,
* hydrops,
* intestinal perforation,
* grade 3 or 4 IVH,
* serum creatinine >1.5,
* previous treatment with a COX inhibitor.

Ages: 1 Minute to 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of PDA Closure | 3 days
  PDA will be evaluated by echocardiography to determined whether it has closed after treatment is complete.

SECONDARY OUTCOMES:
Change in PDA size | 3 days
  Size of PDA will be measured by echocardiography to determine if the size has changed after treatment is complete

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center Neonatal Intesive Care Unit, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No